CLINICAL TRIAL: NCT01441297
Title: A Phase II Study Of BIBF 1120 as Second-line Treatment for Patients With Small Cell Lung Cancer
Brief Title: BIBF 1120 as Second Line Treatment for Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ji-youn Han (Other Government)
Collaborators: National Cancer Center, Korea (Other Government)
Responsible Party: Sponsor-Investigator, Ji-youn Han, Head, Center for Lung Cancer, National Cancer Center, Korea
Organization: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-10-525
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Small Cell Lung Cancer; Small Cell Lung Cancer Recurrent
Keywords: recurrent small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study arm (Experimental): BIBF 1120 study arm
  Interventions: Drug: BIBF 1120

INTERVENTIONS:
Drug: BIBF 1120 — BIBF 1120 200mg bid, PO, daily until PD

SUMMARY:
Although chemotherapy is the primary treatment option for small cell lung cancer (SCLC), longterm survival is rare. SCLC is initially chemosensitive, but rapidly relapses in a chemoresistant form with an overall survival of <5%. Consequently, novel therapies are urgently required and will likely arise from an improved understanding of the disease biology. Some preclinical studies have showed that fibroblast growth factor-2 induces proliferation and

DETAILED DESCRIPTION:
Chemotherapy is the primary treatment option for patients with small cell lung cancer (SCLC), leading to a 5-year survival of about 20% in limited disease (LD), and less than 5% in extensive disease (ED). Although initial tumor response rate to chemotherapy is very high (up to 96% for LD and up to 65% in ED), SCLC relapses in approximately 4 months in ED and 12 months in LD. Despite the administration of second-line chemotherapy, the overall median survival of patients with limited and extensive disease is approximately 18 and 9 months, respectively. In the setting of second-line therapy, response rates to chemotherapy range between 15 and 25%, with median survival in the range of 4-6 months. Second-line therapeutic options include cyclophosphamide, doxorubicin and vincristine (CAV) given every 3 weeks or topotecan, which have similar response rates, time to progression and survival in the two treatment arms (topotecan 24%, 13 and 24.7 weeks; CAV 18%, 12 and 22 weeks, respectively). However, both treatments have substantial toxicities, with 9% of patients on trial withdrawing for toxicity reasons. Treatment-associated mortality was as high as 4.7% (possibly and definitely related), and many patients required transfusion support. Thus, while these treatments have acceptable activity second-line, more active and less toxic treatments are required for this patient population.

The next generation of anti-angiogenic drugs aims to improve clinical efficacy by targeting multiple angiogenic factors. This approach was validated by a recent analysis of BIBF 1120, which inhibits vascular endothelial growth factor receptors (VEGFRs), platelet-derived growth factor receptors (PDGFRs) and the fibroblast growth factor receptors (FGFRs). BIBF 1120 resulted in growth inhibition of tumours in syngeneic rats and human tumour xenografts in nude mice. It also displayed a favourable cellular duration of action and pharmacodynamic profile and was well-tolerated. These data complement early-phase clinical data suggesting that BIBF 1120 might be an effective anti-angiogenic agent. Some preclinical studies have showed that fibroblast growth factor-2 induces proliferation and chemoresistance in SCLC cells. In addition, the selective fibroblast growth factor receptor (FGFR) inhibitor PD173074 blocks H-510 and H-69 SCLC proliferation and clonogenic growth in a dose-dependent fashion and prevents FGF-2-induced chemoresistance. BIBF1120 is a novel, orally available, potent triple angiokinase inhibitor that predominantly blocks the FGFR in addition to vascular endothelial growth factor (VEGF) and platelet-derived growth factor receptor (PDGFR). Therefore, the investigators will conduct a phase II trial to evaluate the efficacy of BIBF1120 in patients with recurrent SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed SCLC
2. Progression during or after prior first line chemotherapy.
3. At least one target tumor lesion RECIST 1.1)
4. Life expectancy of at least three months
5. ECOG PS 0-2
6. Written informed consent

Exclusion Criteria:

1. Previous therapy with other VGFR inhibitors (other than bevacizumab)
2. Persistence of clinically relevant therapy related toxicities from previous chemotherapy and/or radiotherapy
3. Chemo-, hormone-, immunotherapy with monoclonal antibodies, treatment with tyrosine kinase inhibitors, or radiotherapy (except for brain and extremities) within the past 3 weeks prior to treatment with the trial drug i.e., the minimum time elapsed since the last anticancer therapy and the first administration of BIBF 1120 must be 3 weeks
4. Treatment with other investigational drugs or treatment in another clinical trial within the past three weeks before start of therapy or concomitantly with this trial
5. Concomitant yellow fever vaccination
6. Uncontrolled brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease. Patients should have completed surgery or radiation therapy for existing brain metastases, should not have documented increase in size over the previous 3 months and should be asymptomatic off steroids
7. Radiographic evidence of cavitary or necrotic tumors
8. Centrally located tumors with radiographic evidence (CT or MRI) of local invasion of major blood vessels
9. History of clinically significant haemoptysis within the past 3 months (more than one teaspoon of fresh blood per day)
10. Therapeutic anticoagulation (except low dose heparin and/or heparin flush as needed for maintenance of an indwelling intravenous device) or antiplatelet therapy (except for chronic low-dose therapy with acetylsalicylic acid ≤325mg per day)
11. History of major thrombotic or clinically relevant major bleeding event in the past 6 months
12. Known inherited predisposition to bleeding or thrombosis
13. Significant cardiovascular diseases (i.e., hypertension not controlled by medical therapy, unstable angina, history of myocardial infarction within the past 12 months, congestive heart failure > NYHA II, serious cardiac arrhythmia, pericardial effusion)
14. Calculated creatinine clearance by Cockcroft Gault <45ml/min
15. Proteinuria CTCAE grade 2 or greater
16. Total bilirubin above the upper limit of normal
17. ALT and/or AST > 2.5 x upper limit of normal in the presence of live metastasis or ALT and/or AST >1.5 x upper limit of normal in patients without liver metastasis.
18. Prothrombin time and/or partial thromboplastin time greater than 50% deviation from normal limits
19. Platelets <100000 platelets/μL (=mm3)
20. Significant weight loss (> 10 %) within the past 6 weeks prior to treatment in the present trial
21. Current peripheral neuropathy ≥ CTCAE(version4.0) Grade 2 except due to trauma
22. Pre-existing ascites and/or clinically significant pleural effusion
23. Major injuries and/or surgery within the past ten days prior to randomization with incomplete wound healing
24. Serious infections requiring systemic antibiotic (e.g. antiviral, antimicrobial, antifungal) therapy
25. Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
26. Active or chronic hepatitis C and/or B infection
27. Known human immunodeficiency virus (HIV) seropositivity
28. serious illness or concomitant non-oncological disease or
29. Pregnancy or breast feeding
30. Active alcohol or drug abuse
31. Other malignancy within the past three years
32. Hypersensitivity to BIBF 1120 and/or the excipients of the trial drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate | every 8 weeks
  To assess the efficacy of BIBF1120 as second-line treatment in patients with recurrent small cell lung caner

SECONDARY OUTCOMES:
Overall survival rate | every 8 weeks
  Survival time will be calculated from the date of study treatment start to the date of death (or date last seen).
Progression free survival | every 8 weeks
  Progression free survival will be calculated from the date of study treatment start to the first objective documentation of progressive disease or death.
Toxicity | every 4 weeks
  Safety will be evaluated by the frequency, severity, and relationship of adverse events graded by NCI Common Toxicity Criteria (CTC) version 4.0 that occur during the treatment and follow-up periods.

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Youn Han, PhD., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Han JY, Kim HY, Lim KY, Hwangbo B, Lee JS. A phase II study of nintedanib in patients with relapsed small cell lung cancer. Lung Cancer. 2016 Jun;96:108-12. doi: 10.1016/j.lungcan.2016.04.002. Epub 2016 Apr 6. PMID 27133759